CLINICAL TRIAL: NCT07038733
Title: Characterizing the Tumor-draining Lymph Nodes and Other Immune Sites in Renal Cell Carcinoma
Brief Title: Investigation of Lymph Node Biology in Kidney Cancer
Acronym: LN-RCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000039529
Record Dates: First submitted 2025-05-30; First posted 2025-06-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Renal Cell Carcinoma (RCC)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Specimen collection (Experimental): This single arm study will assess adult patients with either a known or suspected kidney cancer referred to Yale Genitourinary Oncology providers in the Yale Urology, Medical Oncology, Radiation Oncology, or Nephrology Departments. Specimens collected will include peripheral blood sample for immune analysis, tumor sample for analysis, adjacent non-malignant kidney for analysis, draining lymph nodes for analysis and finally, regional non-draining lymph nodes for analysis.
  Interventions: Procedure: Peripheral Blood Sample for Immune Analysis; Procedure: Tumor Sample for Analysis; Procedure: Adjacent non-malignant kidney for analysis; Procedure: Draining lymph node(s) for analysis; Procedure: Regional non-draining lymph node(s) for analysis

INTERVENTIONS:
Procedure: Peripheral Blood Sample for Immune Analysis — A peripheral blood sample will be collected at the time of surgery.
Procedure: Tumor Sample for Analysis — Extra tumor which is left over following clinical diagnoses will be collected.
Procedure: Adjacent non-malignant kidney for analysis — Extra normal tissue which is left over following clinical diagnoses will be collected.
Procedure: Draining lymph node(s) for analysis — Draining lymph nodes which have been identified by the surgeon visually, potentially using a tracer (injection of up to 5mg of ICG into the peritumor kidney) will be collected.
Procedure: Regional non-draining lymph node(s) for analysis — Regional lymph nodes which have been deemed as non-draining by the surgeon will be collected.

SUMMARY:
The purpose of this pilot study is to investigate the phenotype, anti-tumor effector functions, and TCR repertoire of T cells isolated from patient tumor draining lymph nodes (TDLNs) to understand T cell priming and trafficking patterns in Renal Cell Carcinoma (RCC). Data and biospecimen collected will be used for current and future research projects involving the study of kidney cancer biology and related medical conditions. We will use this valuable resource to ask clinically relevant translational questions that pertain to biomarker discovery/validation, identification of novel therapeutic targets, and to better understand the genetic and biological basis of the various kidney cancers.

DETAILED DESCRIPTION:
This is a protocol to collect and analyze tissue specimens from patients with kidney cancers. Patients with confirmed or suspected renal cell carcinoma (RCC) evaluated at the YCC Genitourinary Oncology Clinic or participating Smilow Cancer Hospital Care Centers (SCHCC) will be invited to participate in the study.

Participants will consent to the acquisition and analysis of prospective tissue specimens collected at relevant treatment time points (e.g., pre-treatment, response, primary or acquired resistance, and/or at the occurrence of toxicity), based on their cancer treatment course, whether routine care or as part of another clinical trial. Prospective tissue collection include fresh tissue collection at the time of procedures that are conducted at YNHH as part of standard of care (SOC) or clinical trial protocols (procedures billed to either insurance or trial sponsor). Tissue in excess of what is required for diagnostic/clinical uses will be used for research. If an adult participant consents, draining and regional lymph nodes may be obtained for research purposes.

In addition, 20 mL of blood may be collected at time of surgery for correlative biomarker studies and the extraction of germline DNA.

Eligible patients will be identified and consented by their treating clinician (PI or sub- investigators) and/or designated research staff.

ELIGIBILITY:
Inclusion Criteria:

Candidates for inclusion include adult patients with either a known or suspected kidney cancer referred to Yale Genitourinary Oncology providers in the Yale Urology, Medical Oncology and Radiation Oncology or Nephrology Departments. These individuals will be receiving clinical evaluation/medical treatment/surgery/procedures at Yale New Haven Hospital or the Smilow Cancer Hospital.

Participant eligibility will be determined by study investigators and will be offered protocol details. Interested participants will be invited to participate by study investigators. Consent will be obtained by study investigators or other authorized study personnel. Any potential adult participants with known or suspected kidney cancers with a renal mass who are patients of non-study physicians will be invited to participate by study personal only with the approval of their treating physician.

Exclusion Criteria

* Participants under the age of 18. Children will not be enrolled on the study.
* Participants known to be pregnant or actively breastfeeding.
* Iodine allergy hypersensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Molecular Profiling of Tumor and Draining Lymph Node Tissues in Kidney Cancer Patients | 24 months
  This outcome measure focuses on the detailed molecular characterization of tumor and draining lymph node tissues collected from kidney cancer patients. The analysis will include genomic, transcriptomic, and proteomic profiling to understand the underlying biology of kidney cancers
Molecular Responses to Anti-Cancer Therapies in Kidney Cancer Patients | 24 months
  This outcome measure aims to assess the molecular responses of kidney cancer tissues to anti-cancer therapies. It involves analyzing changes in the molecular profiles of tumor and lymph node tissues before and after treatment to evaluate therapeutic efficacy and identify potential biomarkers of response.
Mechanistic Insights into Resistance to Anti-Cancer Therapies in Kidney Cancer | 24 months
  This outcome measure investigates the mechanisms of resistance to anti-cancer therapies in kidney cancer patients. The goal is to identify molecular alterations and signaling pathways associated with resistance, which could inform the development of strategies to overcome or prevent resistance.
Biomarkers for Predicting Toxicities of Anti-Cancer Therapies in Kidney Cancer Patients | 24 months
  This outcome measure aims to identify biomarkers that can predict toxicities associated with anti-cancer therapies in kidney cancer patients. By analyzing molecular changes in tissues, the study seeks to develop predictive models to minimize adverse effects and personalize treatment regimens for better patient management.
  These measures collectively aim to enhance our understanding of kidney cancer biology, responses to therapy, mechanisms of resistance, and toxicity prediction, thereby contributing to more effective and personalized treatment approaches.

CONTACTS AND LOCATIONS:
Overall Officials: David Braun, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No